CLINICAL TRIAL: NCT01381536
Title: GSK1550188, A Randomised, Single-blind, Placebo Controlled, Dose Ascending, Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic of GSK1550188 in Japanese Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Phase I Study of GSK1550188 in Japanese Subjects With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 114243
Record Dates: First submitted 2011-04-21; First posted 2011-06-27 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Anti Blys Antibody
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- GSK1550188 1mg/kg or 10mg/kg (Experimental): one shot IV
  Interventions: Drug: GSK1550188 1mg/kg or 10mg/kg

INTERVENTIONS:
Drug: GSK1550188 1mg/kg or 10mg/kg — IV one shot

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK1550188 in Japanese subjects with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who gave consent to this study participation and signed into informed consent form.
* Subjects who are at least 20 years of age at Screening visit.
* Have a clinical diagnosis of Systemic Lupus Erythematosus (SLE) according to the American College of Rheumatology (ACR) classification criteria, with 4 or more of the 11 ACR criteria present, serially or simultaneously during any interval or observation.
* Be on either no SLE medication or a stable SLE treatment regimen of any medication (e.g., low-dose prednisone, NSAIDs; alone or in combination) for a period of at least 2 months prior to the Screening visit.
* Males and females. A female subject is eligible to enter the study if at least one of the following conditions apply:
* Not pregnant or nursing;
* Of non-childbearing potential (ie, women who had a hysterectomy, are postmenopausal which is defined as 1 year without menses, have both ovaries surgically removed or have current documented tubal ligation); or
* Of childbearing potential (ie, women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea [even severe], women who are perimenopausal or have just begun to menstruate. These women must have a negative serum pregnancy test at screening, and agree to 1 of the following:
* Complete abstinence from penile-vaginal intercourse, when this is the female's preferred and usual lifestyle, from 2 weeks prior to administration of the 1st dose of investigational product until 8 weeks after the last dose of investigational product; or
* Consistent and correct use of 1 of the following acceptable methods of birth control for 1 month prior to the start of the investigational product and for 8 weeks after the last dose of investigational product:
* Implants of etonogestrel or levonorgestrel;
* Estrogenic vaginal ring
* Injectable progesterone
* Any intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
* Oral contraceptives (either combined or progesterone only)
* Double barrier method with vaginal spermicidal agent: Condom and an occlusive cap (cervical cap/vault or diaphragm) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Percutaneous contraceptive patch
* The subject is positive test for anti-nuclear antibody (ANA) or anti-dsDNA antibody in serum

Exclusion Criteria:

* Active lupus nephritis requiring hemodialysis, intravenous cyclophosphamide (Cytoxan),or high-dose prednisone (>60 mg/day) within 6 months prior to the Screening visit
* The subject has severe lupus kidney disease (defined by proteinuria > 6 g/day) within 6 months prior to the Screening visit.
* Received IVIG or plasmapheresis within 6 months prior to Screening visit
* Active CNS lupus [including seizures, psychosis, organic brain syndrome, cerebrovascular accident (CVA), motor neuropathy, vasculitis] requiring medical intervention within 6 months prior to Screening visit
* The subject has hypogammaglobulinemia or IgA deficiency (IgA level < 10 mg/dL)
* History of renal transplant
* History or clinical evidence of active significant acute or chronic diseases (i.e., cardiovascular, pulmonary, untreated hypertension, anemia, gastrointestinal, hepatic, renal, neurological, cancer, or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk
* History of any other medical disease, laboratory abnormalities, or conditions which would make the subject (in the opinion of the Investigator) unsuitable for the study
* History of any infection requiring hospitalization or parenteral antibiotics within 4 weeks prior to Screening visit
* The subject has an abnormality on 12-lead ECG at screening which is clinically significant in the opinion of the investigator.
* The subject is currently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational agent.
* The subject has received a biologic investigational and non-investigational agent within 12 months prior to the dosing day.
* The subject has received a non-biologic investigational agent within 2 months prior to the dosing day.
* Have evidence of current drug or alcohol abuse or dependence.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Have a historically positive HIV test or test positive at screening for HIV.
* History of, or positive test at Screening visit for any of HBsAg, anti-HBcAb or anti-HCVAb. If only anti-HBcAb result is positive, HBV-DNA test will be performed. If HBV-DNA results in negative, the patient is eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07-20 (Actual); Primary Completion 2010-11-27 (Actual); Study Completion 2010-11-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability | For 84 days
  Number of subjects with adverse events (AE) as meaasure of safety and tolerability

SECONDARY OUTCOMES:
To evaluate pharmacokinetics and pharmacodynamics | 84days
  Serum concentrations of GSK1550188 and derived PK parameters for phamacokinetics, Immunoglobulins (IgG, IgM and IgA), complement (C3, C4), CH50, autoantibodies (anti-double stranded deoxyribonucleic acid [dsDNA] and anti-nuclear antibody [ANA]), B cell subsets (CD20+, CD20+/27+ memory, CD20+/27-naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells), anti-belimumab antibody, BLyS protein, and Safety of Estrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) score

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Miyagi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Yamada M, Akita M, Nakagawa T, Takahashi N, Endo A, Yoshida P. Safety, tolerability, pharmacokinetics and pharmacodynamics of belimumab in Japanese patients with mild-to-moderate systemic lupus erythematosus. J Drug Assess. 2013 Apr 12;2(1):40-8. doi: 10.3109/21556660.2013.792823. eCollection 2013. PMID 27536436
- See also: Results for study 114243 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114243?search=study&search_terms=114243#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 114243 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114243 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114243 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114243 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114243 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114243 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register